CLINICAL TRIAL: NCT04833348
Title: Quantification of Motor Function in Infants With Spinal Muscular Atrophy Treated With Innovative Therapies, IMUSMA Project
Brief Title: Quantification of Motor Function in Infants With Spinal Muscular Atrophy Treated With Innovative Therapies
Acronym: IMUSMA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP201640; 2020-A02279-30 (Other: ID-RCB Number)
Record Dates: First submitted 2021-03-23; First posted 2021-04-06 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal muscular atrophy; Innovative therapies; Motor function; Wearable inertial sensors
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): Infants with spinal muscular atrophy cared by the Neuromuscular Reference Center at Necker Hospital and eligible for innovative therapy (gene therapy or pharmacogenetics)
  Interventions: Other: Motor function measurement using inertial sensors

INTERVENTIONS:
Other: Motor function measurement using inertial sensors — Measurement of motor skills at M0: start of the administration of the innovative therapy and then 1 month, 3 months, 6 months, 1 year and then 2 years later:
  * Free motor skills in the supine position
  * Motricity in the supine position stimulated by a play frame
  * Measurement of the proximal and distal activity of the upper limbs in motor skills stimulated by the play gantry
  * Measurement of activity in a supported sitting position Longitudinal study, the subject is his own control

SUMMARY:
The aim of the study is to propose a method for quantifying motor function in infants with spinal muscular atrophy treated with innovative therapies using inertial sensors.

DETAILED DESCRIPTION:
Infantile spinal muscular atrophy is a common disease (the second most common fatal autosomal recessive disease after cystic fibrosis), neurodegenerative disorders of childhood causing severe motor impairment and a risk to life through respiratory failure in the most severe forms.

Innovative therapies (gene therapy or pharmacogenetics) have recently proven their effectiveness on survival criteria. Nevertheless, the motor benefit of these therapies must be evaluated more precisely.

Currently, the reference methods for motor development assessment are fairly robust semi-quantitative motor scales that lack sensitivity and do not reflect function (CHOPINTEND, HINE, BAYLEY SCALE, MFM and CGI-scale).

Advances in recent techniques have enabled the emergence of non-invasive, secure, easy-to-use inertial sensors in routine clinical practice that allow quantification of infant movements.

The aim of the study is to propose a method for quantifying motor function in infants with spinal muscular atrophy treated with innovative therapies using inertial sensors.

ELIGIBILITY:
Inclusion Criteria:

* Infants of both sexes
* Suffering from spinal muscular atrophy (diagnosis by genetic study "homozygous deletion of SMN1")
* Followed up by the Necker Neuromuscular Reference Center (GNMH)
* Eligible for innovative therapy (gene therapy or pharmacogenetics)

  * age of onset of the disease <1 year
  * no severe respiratory impairment (dependence on ventilatory support for more than 16 hours per day) or bulbar involvement
  * decision of treatment by a Multidisciplinary Consultation Meeting national of experts
* Benefiting from social security scheme
* Informed consent signed by holders of parental authority and the investigator

Exclusion Criteria:

* Non-consent of one of the holders of parental authority
* Respiratory instability (dependence on ventilatory support for more than 16 hours per day) or hemodynamics
* Contraindication to innovative therapy
* History of another disease impacting motor skills (neonatal suffering, etc.)

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in the 95th percentile of the norm of acceleration | Month 0 to month 24
  95th percentile of the norm of the acceleration of the feet and the arms.

SECONDARY OUTCOMES:
Change in the 95th percentile of the norm of angular velocity | Month 0 to month 24
  95th percentile of the norm of angular velocity of the feet and the arms.
Change in the 95th percentile of the accelerations allong the vertical axis and the horizontal plane | Month 0 to month 24
  95th percentile of the accelerations of the feet and the arms the vertical axis and the horizontal plane.
Change in the 95th percentile of the angular velocities allong the vertical axis and the horizontal plane. | Month 0 to month 24
  95th percentile of the angular velocities of the feet and the arms the vertical axis and the horizontal plane.
Change in the acceleration's entropy | Month 0 to month 24
  Acceleration's entropy computed in the different axis of the feet and the arms.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle DESGUERRE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Brian TERVIL, PhD, Study Director — Centre Borelli - Université Paris Descartes
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No